CLINICAL TRIAL: NCT06032091
Title: Digital Phenotyping for Changes in Activity at the End of Life in People With Dementia: an Observational Trial Based on Sensing Technology
Brief Title: Digital Phenotyping for Changes in Activity at the End of Life in People With Dementia
Acronym: DIPHDEM
Status: Recruiting | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Helse Vest (Other); Haukeland University Hospital (Other); Haraldsplass Deaconess Hospital (Other); Bergen Red Cross Nursing Home (Unknown)
Responsible Party: Sponsor
Other Study IDs: F-12829-D10484
Record Dates: First submitted 2023-06-09; First posted 2023-09-11 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-10

CONDITIONS: Dementia
Keywords: end-of-life care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Persons with dementia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The study is observational and will not include any specific interventions other than the regular care practice that the participants receive from their care providers. The study will use a wrist-mounted smartwatch for monitoring. Previous studies show acceptability toward wearable devices among persons with dementia; however, if the care staff recognize discomfort or distress caused by the device, it will be immediately removed.

SUMMARY:
Background:

Almost 90% of people with dementia develop serious symptoms such as apathy, agitation, pain, and sleep disturbances. Movement and participation in daily activities also decrease dramatically over time. Traditional measures for these symptoms are usually in the form of a questionnaire and are not very accurate. Technology, such as a smartwatch, can be an effective tool for complementing traditional measures. Currently, there are few studies which look at activity and symptom measurements at the end-of-life. This makes results from this study extremely valuable for future care decisions, especially for people which may not be able to communicate their needs during the end-of-life period.

Method/Design:

DIgital PHenotyping in DEMentia (DIPH.DEM), a 3-year cross-sectional observational study (N=50), will look at activities, apathy, agitation, and sleep disturbances using sensing technologies to monitor participants at the end of life. The objective of the study is to use a smartwatch and wireless radar (bedside) device (Somnofy), in addition to validated assessment tools to describe the activity patterns for patients with dementia at the end of life (baseline and every 6.months). We hypothesize that this will enable better estimation of time of death, facilitating discussion surrounding improvement of end-of-life interventions and directives.

Discussion:

The use of sensors (smartwatch and wireless beside device) can provide valuable knowledge on living and dying with dementia, improve end-of-life directives, and provide guidance for timely, appropriate interventions, including referral to palliative services.

Impact on society:

DIPH.DEM has the potential to enable more timely, precise, and quality care for people with dementia living at home, in nursing homes, and hospitals.

DETAILED DESCRIPTION:
About 90% of people with dementia develop behavioral and psychological symptoms such as agitation, depression and psychosis. In addition, their activity levels decrease over time. Traditional outcome measures can capture physical, mental and social activities of clinical conditions, but usually have low validity. The use of sensor technology in people with dementia is currently poorly validated. DIPH.DEM will examine whether digital tools such as a smartwatch and Somnofy (radar installation) can provide objective measurements of the patient's activities and symptoms throughout the nursing home/hospital stay, including the end of life phase. The participants are people with dementia, >64 years, who are living in a nursing home. A selection of traditional tools and sensor data is collected at baseline and every 6 months (7 days continuous monitoring). If the participant has a significant change in health status, we will begin with continuous sensor measurements until the end of life (up to 12 weeks). DIPH.DEM can provide valuable information on activity development and symptom presentation toward the end of life in people with dementia. Informal caregivers (usually a family member) will be included to assist with the outcome measures within the study. Participants will be recruited from the Health Region West Norway and Bergen Municipality (sampling method is by invitation to volunteer). All consent procedures will be developed in accordance with Norwegian law.

ELIGIBILITY:
Inclusion Criteria:

* People with dementia or who have a likely diagnosis of dementia
* Hospital (admitted for >3 days)
* Nursing home resident
* >64 years old
* Score of <4 on the 4 A's Test for Delirium (4AT) will be required for inclusion (no delirium)

Exclusion Criteria:

* People without dementia or cognitive impairment
* People that are considered already in a health status emergency (< 6 weeks to live)
* People that are not living in the nursing home

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults with dementia or cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Activities of Daily Living (ADL) - Physical Self Maintenance Scale (PSMS), Lawton and Brody, 1969. | Baseline and every 6.months (up to one year)
  Personal functional daily activities such as toileting, eating, self-care, movement/ambulation, transfers, bathing. 6 sections - scoring 1-5 on each, higher score indicates greater disability.
Digital biomarker estimations for apathy, agitation, pain, and sleep disturbances | Baseline and every 6.months (up to one year), continuous up to 12 weeks if a serious health event occurs
  Estimation of activity changes and selected behavioral disturbances resulting from the combined digital phenotype modeling; these estimations are experimental and "scores" will be based on analysis of found data after data collection period.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory - Nursing Home Version (NPI-NH) | Baseline and every 6.months (up to one year)
  Validated in Norwegian nursing homes, measuring symptoms of behavioral and psychological symptoms of dementia (BPSD) such as: apathy, agitation, depression, anxiety, sleep disturbance, and appetite/eating. Gives scores 1-4 (higher numbers being daily occurance) for amount, 1-3 for intensity and burden of care related to symptom for caregiver (1-5) for each symptom.
Mobilization, Observation, Behavioral, Intensity Dementia (MOBID-2) | Baseline and every 6.months (up to one year)
  Measurement of pain specific to a dementia population; visual analog scale alongside likert scale 0-10, 0 being no pain and 10 being the worst pain, validated with persons with dementia
InterRai-Palliative Care (InterRai-PC) | Baseline and every 6.months (up to one year)
  Oral health section only/specific of the InterRai-PC, assessment of symptoms
Digital secondary outcomes | Baseline and every 6.months (up to one year)
  Device-native scores for activity and sleep.
Edmonton Symptom Assessment System (ESAS++) | Baseline and every 6.months (up to one year)
  Symptom assessment for palliative care period and the end of life period, with added items: death rattle, dyspnea, sleep disturbances, emesis specific to end of life. Likert scale 0-10; 0 indicating no symptoms and 10 is worst symptom.

OTHER OUTCOMES:
Chart review | Baseline
  A medication list will be compiled according to the Anatomical Therapeutic Chemical classification (ATC codes) and the Defined Daily Dose (DDD) of regularly scheduled treatments.
Clinical Dementia Rating (CDR) | Baseline
  Classification of cognitive impairment, 0 no cognitive impairment, 0.5 questionable impairment, 1 mild cognitive impairment, 2 moderate cognitive impairment, 3 severe cognitive impairment.
General Medical Health Rating Scale (GMHR) | Baseline
  Mortality risk measure for general wellbeing, medical comorbidity, degree of somatic illness; top 2 scores are good, bottom 2 indicate serious illness with comorbidities. Bedside measure validated in NH with people with dementia.
4 A's Test for Delirium (4AT) | Baseline
  Distinction between dementia and delirium for inclusion to study, >4 indicates delirium; will be used as an exclusion criteria (particpants must score <4)
Clinical Frailty Scale (CFS) | Baseline
  Mortality risk measure for general wellbeing, higher scores indicate greater disability (1-9)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina S Husebo, MD, PhD, Study Director — University of Bergen, Center for Elderly and Nursing Home Medicine, Neuro-SysMed Center; Monica Patrascu, Eng, PhD, Principal Investigator — University of Bergen, Center for Elderly and Nursing Home Medicine, Neuro-SysMed Center; Lydia Boyle, MSc, DPT, Study Chair — University of Bergen, Center for Elderly and Nursing Home Medicine, Neuro-SysMed Center
Locations (1):
- Bergen Røde Kors Sykehjem AS, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Based on previous experience, more data is often produced than is used in a single PhD project. This also applies to data that can be viewed and analyzed in a new context. In recent years, we have had good experience in using existing data for new PhD candidates (such as the first article in the course of the PhD studies) or for collaboration partners who send Master students/PhD candidates to our center to carry out new analyses. This may include data from traditional outcome measures or sensor data. The University of Bergen will always retain management rights and only share anonymized data for local use.

REFERENCES:
- [Background] Sallnow L, Smith R, Ahmedzai SH, Bhadelia A, Chamberlain C, Cong Y, Doble B, Dullie L, Durie R, Finkelstein EA, Guglani S, Hodson M, Husebo BS, Kellehear A, Kitzinger C, Knaul FM, Murray SA, Neuberger J, O'Mahony S, Rajagopal MR, Russell S, Sase E, Sleeman KE, Solomon S, Taylor R, Tutu van Furth M, Wyatt K; Lancet Commission on the Value of Death. Report of the Lancet Commission on the Value of Death: bringing death back into life. Lancet. 2022 Feb 26;399(10327):837-884. doi: 10.1016/S0140-6736(21)02314-X. Epub 2022 Feb 1. No abstract available. PMID 35114146
- [Background] Sandvik RK, Selbaek G, Bergh S, Aarsland D, Husebo BS. Signs of Imminent Dying and Change in Symptom Intensity During Pharmacological Treatment in Dying Nursing Home Patients: A Prospective Trajectory Study. J Am Med Dir Assoc. 2016 Sep 1;17(9):821-7. doi: 10.1016/j.jamda.2016.05.006. Epub 2016 Jun 16. PMID 27321869
- [Background] Abbott KM, Bangerter LR, Humes S, Klumpp R, Van Haitsma K. "It's important, but...": Perceived Barriers and Situational Dependencies to Social Contact Preferences of Nursing Home Residents. Gerontologist. 2018 Nov 3;58(6):1126-1135. doi: 10.1093/geront/gnx109. PMID 28645167
- [Background] Vik-Mo AO, Giil LM, Borda MG, Ballard C, Aarsland D. The individual course of neuropsychiatric symptoms in people with Alzheimer's and Lewy body dementia: 12-year longitudinal cohort study. Br J Psychiatry. 2020 Jan;216(1):43-48. doi: 10.1192/bjp.2019.195. PMID 31506117
- [Background] Faeo SE, Husebo BS, Bruvik FK, Tranvag O. "We live as good a life as we can, in the situation we're in" - the significance of the home as perceived by persons with dementia. BMC Geriatr. 2019 Jun 6;19(1):158. doi: 10.1186/s12877-019-1171-6. PMID 31170916
- [Background] Husebo BS, Heintz HL, Berge LI, Owoyemi P, Rahman AT, Vahia IV. Sensing Technology to Monitor Behavioral and Psychological Symptoms and to Assess Treatment Response in People With Dementia. A Systematic Review. Front Pharmacol. 2020 Feb 4;10:1699. doi: 10.3389/fphar.2019.01699. eCollection 2019. PMID 32116687
- [Background] Vahia IV, Forester BP. Motion mapping in humans as a biomarker for psychiatric disorders. Neuropsychopharmacology. 2019 Jan;44(1):231-232. doi: 10.1038/s41386-018-0205-7. No abstract available. PMID 30214060
- [Background] Au-Yeung WM, Miller L, Beattie Z, May R, Cray HV, Kabelac Z, Katabi D, Kaye J, Vahia IV. Monitoring Behaviors of Patients With Late-Stage Dementia Using Passive Environmental Sensing Approaches: A Case Series. Am J Geriatr Psychiatry. 2022 Jan;30(1):1-11. doi: 10.1016/j.jagp.2021.04.008. Epub 2021 Apr 22. PMID 34039534
- [Background] Torrado JC, Husebo BS, Allore HG, Erdal A, Faeo SE, Reithe H, Forsund E, Tzoulis C, Patrascu M. Digital phenotyping by wearable-driven artificial intelligence in older adults and people with Parkinson's disease: Protocol of the mixed method, cyclic ActiveAgeing study. PLoS One. 2022 Oct 14;17(10):e0275747. doi: 10.1371/journal.pone.0275747. eCollection 2022. PMID 36240173
- [Background] Schuurmans AAT, de Looff P, Nijhof KS, Rosada C, Scholte RHJ, Popma A, Otten R. Validity of the Empatica E4 Wristband to Measure Heart Rate Variability (HRV) Parameters: a Comparison to Electrocardiography (ECG). J Med Syst. 2020 Sep 23;44(11):190. doi: 10.1007/s10916-020-01648-w. PMID 32965570
- [Background] Toften S, Pallesen S, Hrozanova M, Moen F, Gronli J. Validation of sleep stage classification using non-contact radar technology and machine learning (Somnofy(R)). Sleep Med. 2020 Nov;75:54-61. doi: 10.1016/j.sleep.2020.02.022. Epub 2020 Mar 6. PMID 32853919
- [Background] Jorm AF. The Informant Questionnaire on cognitive decline in the elderly (IQCODE): a review. Int Psychogeriatr. 2004 Sep;16(3):275-93. doi: 10.1017/s1041610204000390. PMID 15559753
- [Background] Reisberg B. Functional assessment staging (FAST). Psychopharmacol Bull. 1988;24(4):653-9. No abstract available. PMID 3249767
- [Background] Evensen S, Hylen Ranhoff A, Lydersen S, Saltvedt I. The delirium screening tool 4AT in routine clinical practice: prediction of mortality, sensitivity and specificity. Eur Geriatr Med. 2021 Aug;12(4):793-800. doi: 10.1007/s41999-021-00489-1. Epub 2021 Apr 4. PMID 33813725
- [Background] Thorpe O, McCabe E, Herrero EM, Doyle WO, Dillon A, Edge L, Flynn S, Mullen A, Davis A, Molamphy A, Kirwan A, Briggs R, Lavan AH, Shields D, McMahon G, Hennessy A, Kennedy U, Staunton P, Kidney E, Yeung SJ, Glynn D, Horgan F, Cunningham C, Romero-Ortuno R. Scoring the Clinical Frailty Scale in the Emergency Department: The Home FIRsT Experience. J Frailty Sarcopenia Falls. 2022 Jun 1;7(2):95-100. doi: 10.22540/JFSF-07-095. eCollection 2022 Jun. PMID 35775090
- [Background] Lyketsos CG, Galik E, Steele C, Steinberg M, Rosenblatt A, Warren A, Sheppard JM, Baker A, Brandt J. The General Medical Health Rating: a bedside global rating of medical comorbidity in patients with dementia. J Am Geriatr Soc. 1999 Apr;47(4):487-91. doi: 10.1111/j.1532-5415.1999.tb07245.x. PMID 10203127
- [Background] Hui D, Bruera E. The Edmonton Symptom Assessment System 25 Years Later: Past, Present, and Future Developments. J Pain Symptom Manage. 2017 Mar;53(3):630-643. doi: 10.1016/j.jpainsymman.2016.10.370. Epub 2016 Dec 29. PMID 28042071
- [Background] Selbaek G, Kirkevold O, Sommer OH, Engedal K. The reliability and validity of the Norwegian version of the Neuropsychiatric Inventory, nursing home version (NPI-NH). Int Psychogeriatr. 2008 Apr;20(2):375-82. doi: 10.1017/S1041610207005601. Epub 2007 Jun 11. PMID 17559707
- [Background] Husebo BS, Ostelo R, Strand LI. The MOBID-2 pain scale: reliability and responsiveness to pain in patients with dementia. Eur J Pain. 2014 Nov;18(10):1419-30. doi: 10.1002/ejp.507. Epub 2014 May 5. PMID 24799157
- [Background] Park C, Mishra R, Golledge J, Najafi B. Digital Biomarkers of Physical Frailty and Frailty Phenotypes Using Sensor-Based Physical Activity and Machine Learning. Sensors (Basel). 2021 Aug 5;21(16):5289. doi: 10.3390/s21165289. PMID 34450734
- [Background] Browne B, Kupeli N, Moore KJ, Sampson EL, Davies N. Defining end of life in dementia: A systematic review. Palliat Med. 2021 Dec;35(10):1733-1746. doi: 10.1177/02692163211025457. Epub 2021 Jun 17. PMID 34137314
- [Background] Taylor-Rowan M, Nafisi S, Owen R, Duffy R, Patel A, Burton JK, Quinn TJ. Informant-based screening tools for dementia: an overview of systematic reviews. Psychol Med. 2023 Jan;53(2):580-589. doi: 10.1017/S0033291721002002. Epub 2021 May 25. PMID 34030753
- [Background] Puaschitz NG, Jacobsen FF, Mannseth J, Angeles RC, Berge LI, Gedde MH, Husebo BS. Factors associated with access to assistive technology and telecare in home-dwelling people with dementia: baseline data from the LIVE@Home.Path trial. BMC Med Inform Decis Mak. 2021 Sep 15;21(1):264. doi: 10.1186/s12911-021-01627-2. PMID 34525979
- [Background] Johansen RH, Olsen K, Bergh S, Benth JS, Selbaek G, Helvik AS. Course of activities of daily living in nursing home residents with dementia from admission to 36-month follow-up. BMC Geriatr. 2020 Nov 20;20(1):488. doi: 10.1186/s12877-020-01877-1. PMID 33218298